CLINICAL TRIAL: NCT03330886
Title: An Observational Study of the Safety of Atezolizumab in Patients With Advanced or Metastatic Urothelial Carcinoma in Argentina
Brief Title: A Study of the Safety of Atezolizumab in Patients With Advanced or Metastatic Urothelial Carcinoma in Argentina
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML39853
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered via IV at a 1200-mg dose over 60 minutes every 3 weeks (to be reduced to 30 minutes every 3 weeks if the first dose is tolerated).

SUMMARY:
The main purpose is to study the safety and effectiveness of atezolizumab in patients with locally advanced or metastatic urothelial carcinoma whose disease has worsened during or following platinum-containing chemotherapy, or within 12 months of receiving platinum-containing chemotherapy, either before (neoadjuvant) or after (adjuvant) surgical treatment in common clinical practice settings in Argentina.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent form submitted to the Administración Nacional de Medicamentos Alimentos y Tecnología Médica (ANMAT)
* Histologically or cytologically documented locally advanced or metastatic urothelial carcinoma (including renal pelvis, ureters, urinary bladder, and urethra).
* Have received at least one dose of atezolizumab as per local label and clinical practice.

Exclusion Criteria:

* Contraindicated atezolizumab therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically or cytologically documented locally advanced or metastatic urothelial carcinoma (including renal pelvis, ureters, urinary bladder, and urethra) that have received the indication for treatment with atezolizumab as per local label (disease progression during or following platinum containing therapy) in the context of routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AE) | Up to approximately 2 years.

SECONDARY OUTCOMES:
Percentage of participants with Confirmed Objective Response (ORR) of Complete Response (CR) or Partial Response (PR) | Up to approximately 2 years.
Duration of Response (DOR) | Up to approximately 2 years.
Progression Free Survival (PFS) | Up to approximately 2 years.
Overall Survival (OS) | Up to approximately 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Productos Roche S.A. Quimica e Industrial, División Farmacéutica, Buenos Aires, Argentina